CLINICAL TRIAL: NCT02362529
Title: Biomarkers of Neuroinflammation and Anti-Inflammatory Treatments in Major Depressive Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Head Neurochemical Imaging in Mood Disorders, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REB056/2014
Record Dates: First submitted 2015-02-04; First posted 2015-02-13 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Minocycline; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Minocycline (Experimental): The dose of minocycline would be 50mg per day on week 1, 50mg bid on week 2 and 100mg bid weeks 3-8. For tapering, the dose will be reduced to 50mg bid for a week, and then stopped.
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): The number and appearance of the pills would be identical to those in the minocycline arm.
  Interventions: Drug: Placebo
- Celecoxib (Other): This will be an open label trial for those with Hamilton Depression Rating Scale score ≥ 8 following the minocycline v. placebo trial or those not eligible for Phase 2. Dose of celecoxib will be 100 mg bid for the first week and 200mg bid for weeks 2-8. For tapering, the dose of celecoxib will be reduced to 100mg bid for one week, and then stopped.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Minocycline — 50 mg and 100 mg capsule, oral administration
  Other Names: Mylan-minocycline
  Arms: Minocycline
Drug: Placebo — Lactose monohydrate in identical gel capsules to minocycline, oral administration.
  Other Names: Lactose monohydrate
  Arms: Placebo
Drug: Celecoxib — 100 mg and 200 mg capsules, oral administration.
  Other Names: Celebrex (Pfizer)
  Arms: Celecoxib

SUMMARY:
The purpose of this study is to determine if translocator protein total distribution volume (TSPO VT) is elevated in major depressive disorder that is not responding to medication and if adding minocycline can affect TSPO VT. Many remain treatment resistant with common antidepressant treatments and the investigators think it may be due to poor targeting of brain pathologies.

DETAILED DESCRIPTION:
There will be three Phases in the study. Only MDE subjects will be invited to continue to Phase 2 and 3. Subjects will be invited to continue to the subsequent Phase given they meet entry criteria described below:

Phase 1: The investigators will evaluate whether TSPO is elevated in individuals during a current MDE compared to healthy controls. Eligible participants will receive one [18F]FEPPA PET scan and one MRI scan. Other measures will include urine sample, blood samples for genetic and peripheral biomarker analysis, a neurocognitive battery, mood scales and questionnaires.

Phase 2: Participants who have elevated TSPO VT in Phase 1 and are agreeable to receiving minocycline will be invited to participate in Phase 2. Based on our previous results participants will be considered candidates for Phase 2 if TSPO VT ≥ 10.5 (HAB) or ≥8.5 (MAB) in any of the primary regions of interest (prefrontal cortex, anterior cingulate cortex or insula). Eligible participants will be invited to participate in a randomized, double blind, placebo controlled trial, to receive either minocycline or placebo. After the eight weeks of treatment, participants will receive one [18F]FEPPA PET scan. Other measures will include urine samples, blood samples, mood scales and questionnaires.

Phase 3: If, after the initial eight week treatment period with either minocycline or placebo, any participant continues to have depressive symptoms (17-item Hamilton Depression Rating Scale score ≥ 8) they will be invited to participate in an eight week open label trial of celecoxib. Participants not eligible for Phase 2 may also be invited to participate in Phase 3 directly from Phase 1.

ELIGIBILITY:
Group 1 - Current major depressive episode (MDE) secondary to MDD

Inclusion Criteria:

* good physical health with no active medical conditions
* non-cigarette smoking
* no past or current substance abuse or dependence
* negative urine pregnancy test at screening and scan days (for women)
* primary diagnosis of current major depressive episode (MDE) and major depressive disorder (MDD) verified by SCID for DSM IV
* score greater than 19 on the 17 item HDRS
* non-response to a clinical trial of at least one antidepressant given at appropriate clinical dose
* willing to take medication for the duration of the trial and has previously taken antidepressants for the duration of the trial
* presently taking an antidepressant at a standard clinical dose.

Exclusion Criteria:

* history of neurological illness or autoimmune disorders
* never taken a tricyclic antidepressant or an antidepressant that raises norepinephrine
* received treatment with electroconvulsive therapy or mechanical brain stimulation in the previous 6 months
* currently taking medication contraindicated or that may possibly interact with either minocycline or celecoxib
* known intolerance or allergy to minocycline, other tetracyclines, sulfonamides or NSAIDs
* taken diazepam or other benzodiazepine use within the past month, except for lorazepam and clonazepam
* use of anti-inflammatory drugs or tetracyclines lasting ≥1 week within the past month
* history of severe hepatic or renal insufficiency, asthma, allergies, gastrointestinal disease, ischemic heart disease, cerebrovascular disease or congestive heart failure
* lactose intolerance

Group 2 - Healthy Controls - Phase 1 (baseline scan) only

Inclusion criteria:

* score below 8 on the 17 item HDRS
* good physical health
* non-cigarette smoking
* negative urine pregnancy test at screening and scan days (for women)
* negative urine screen for drugs of abuse

Exclusion criteria:

* past or current diagnosis of axis I or axis II disorder as determined by the SCID I and SCID II for DSM IV
* history of psychotropic medication use
* history of neurological illness or autoimmune disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Translocator total distribution volume (TSPO VT): Treatment Effect of Minocycline in MDE Subjects | Pre- and post-minocycline or placebo treatment= 8 weeks total between pretreatment and posttreatment scans
  TSPO VT will be measured using [18F]FEPPA positron emission tomography brain scans. Eligible MDE participants will be randomized to either minocycline or placebo. Following 8 weeks of either minocycline or placebo treatment, MDE participants will have a second PET scan .
Translocator total distribution volume (TSPO VT): Difference between MDE and healthy subjects | Pre-treatment scan will take place up to 8 weeks from initial assessment
  Compare baseline TSPO VT prior to treatment between MDE group and healthy group

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale Score | Pre- and post-minocycline treatment (8 weeks total between pre- and post-treatment). Pre- and post-celecoxib treatment (8 weeks total between pre- and post-treatment).
  Change in HDRS score following minocycline vs. placebo treatment. Change in HDRS score following celecoxib treatment.

OTHER OUTCOMES:
Hopkins Verbal Learning Test-Revised | Pre- and post-minocycline or placebo treatment (8 weeks between pre- and post-treatment measure)
  To assess verbal memory we will administer the Hopkins Verbal Learning Test-Revised to MDE participants before and after treatment.
Brief Visuospatial Memory Test-Revised | Pre- and post-minocycline or placebo treatment (8 weeks between pre- and post-treatment measure)
  To assess visuospatial memory we will administer the Brief Visuospatial Memory Test-Revised to MDE participants before and after treatment.
Comprehensive Trails Making Test | Pre- and post-minocycline or placebo treatment.
  To assess psychomotor speed and attention we will administer the Comprehensive Trails Making Test to MDE participants before and after treatment.
Genetic sample | Phase 1-single sample
  The priority of the genetic sample is to analyze the alleles of polymorphism rs6971 which has an association with the affinity of most second generation TSPO ligands including [18F]FEPPA. The genetic sample will also be used to study sequences of genes that are believed to affect TSPO expression, inflammation, mood and conditions that may predispose to mood disorders.
Blood samples (serum and plasma) | Pre- and post-minocycline or placebo treatment (8 weeks between measures). Pre- and post-celecoxib treatment (8 weeks between measures).
  Analyses will include complete blood cell count (CBC), ESR, hepatic and renal function. Peripheral marker analyses will include proteins related to TSPO expression and inflammation. Plasma minocycline and celecoxib levels will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health; University of Toronto
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada